CLINICAL TRIAL: NCT04292132
Title: Prospektive Langzeitstudie Zur Implantatprothetischen Versorgung
Brief Title: Two Interforaminal Implants in an Immediate or Delayed Loading Protocol for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Neoss Ltd., Harrogate, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUGraz Neoss1
Record Dates: First submitted 2019-06-26; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Edentulous Jaw
Keywords: Dentistry; Mandibular Atrophy; Mandibular Overdenture
MeSH Terms: conditions — Jaw, Edentulous | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional loading (Active Comparator): Loading of 4 interforaminal implants three months after surgery.
  Interventions: Procedure: Implant placement; Procedure: conventional loading
- Immediate Loading (Experimental): Loading of 4 interforaminal implants immediately after surgery.
  Interventions: Procedure: Implant placement; Procedure: immediate loading

INTERVENTIONS:
Procedure: Implant placement — interforaminal placement of 2 implants
Procedure: immediate loading — immediate loading with a locator retained mandibular overdenture
  Arms: Immediate Loading
Procedure: conventional loading — conventional loading with a locator retained mandibular overdenture 3 months postoperatively
  Arms: Conventional loading

SUMMARY:
The study population comprises 20 completely edentulous patients aged 60 years and older with severe mandible resorption. Each patient receives two inter-foraminal implants (Neoss Ltd., Harrogate, UK). Following randomization, implants are loaded either immediately after dental implant surgery or three months after implant placement with the Locator®-abutment system. At follow-up visits 3, 6 12, 24 and 36 months after loading, implant stability is evaluated with Periotest® and Ostell®.

DETAILED DESCRIPTION:
Hypothesis:

Especially for gerontoprosthetics, the Locator® abutment system offers the possibility of a minimally invasive retention of prosthetic total restorations of edentulous mandibles. The reduced number of 2 interforaminal implants is intended to ensure implantological anchoring with minimal surgical, technical, financial and time expenditure.

Research Question:

How safe is this minimally invasive and cost-effective implant and anchoring system in terms of long-term outcome? Are the two implant-prosthetic procedures (immediate versus late restoration) different in terms of implant survival time?

Materials and methods

Enrollment:

* 20 patients without relevant pre-existing conditions, from the age of 60 years
* edentulous mandible, alveolar ridge atrophy

Statistical Analysis:

When planning the study, it is estimated that bone resorption in the peri-implant area of the immediate-care implants is greater than in the late-treated implants. 10 patients per group are required with a t-test (α = 0.05) and a power of 80% if the null hypothesis is formulated as follows: -difference of means is 0 and the alternative - expected difference of means is 1mm, common standard deviation is 0.75.

Collective A (open healing - immediate loading): Insertion of a new, prefabricated total mandibular prosthesis on the day of the operation immediately postoperatively after screwing in the Locator® abutments.

Polymerization of the corresponding Locator® matrices in the newly incorporated lower jaw denture in the patient's mouth.

Collective B (closed implant healing - conventional loading): 3 months after implantation Exposure of the primary closed implants. Immediately following insertion of the prefabricated full-thickness UK prosthesis and retention by the implants using Locator® abutments.

Test parameters:

1. Intraoperative torque measurement in Ncm
2. Radiological measurement of periimplant bone height using orthopantomogram
3. 4-point measurement of peri-implant probing depth using WHO periodontal probe. The measurement is mesial, distal, buccal and lingual of the implant.
4. Measurement of bleeding on probing (parameters of peri-implant inflammation) using the WHO periodontal probe.
5. Analysis of implant stability using the Periotest® and Osstell® measuring instruments according to a standardized scheme: The strength values are performed in a measuring range consisting of a straight line through the center of the implant and the resulting 180 ° circle sector anterior to this line results. After multiple measurements (5-fold) the lowest numerical value for the Periotest® and for the RFA (Osstell®) the lowest value documented.

ELIGIBILITY:
Inclusion Criteria:

* 60 or older
* edentulous lower jaw with advanced atrophy
* poor fit and retention even with a new prosthesis

Exclusion Criteria:

* poor general condition (ASA classification grade IV or more), or
* high risk situations for implant therapy (e.g. disorders of bone metabolism due to antiresorptive therapy)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Implant stability | 0,3,6,12,24,36 months
  Evaluation of Implant stability with Resonance frequency analysis (Ostell®) indicating quality of osseointegration
Change of Implant stability | 0,3,6,12,24,36 months
  Evaluation of implant stability with electromechanical tapping (Periotest®) indicating quality of osseointegration

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Acham, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No